CLINICAL TRIAL: NCT07182877
Title: A Randomized Controlled Trial to Compare the Dwell Time of Open and Closed-type Peripheral Catheters in Patients Admitted to the Respiratory Intensive Care Unit
Brief Title: Comparison of Dwell Time of Open Versus Closed Type Peripheral Intravenous Cannula
Acronym: COT-cannula
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC-INT/2024/Study-2393
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Comparison of Dwell Time of Two Different Types of Intravenous Cannula
Keywords: IV cannula, thrombophlebitis
MeSH Terms: conditions — Thrombophlebitis

STUDY DESIGN:
Intervention Model Description: Group 1: closed-type peripheral catheters Group 2: open-type peripheral catheters
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Closed-type peripheral catheters
  Interventions: Device: Closed-type peripheral cannula
- Group 2 (Active Comparator): Open-type peripheral catheters
  Interventions: Device: Open type peripheral cannula

INTERVENTIONS:
Device: Closed-type peripheral cannula — We will use closed-type peripheral catheters (BD Nexia Closed IV Catheter System.
  Other Names: Closed cannula
  Arms: Group 1
Device: Open type peripheral cannula — We will use POLYMED Ultra Intravenous cannula in the control arm
  Other Names: Open cannula
  Arms: Group 2

SUMMARY:
Studies have shown that stabilisation devices are associated with fewer complications and lower failure rates in peripheral catheters.3,6,7 Although closed-system peripheral catheters offer potential advantages, such as reduced manipulation of components and minimised blood spillage, more research is needed to understand their impact on outcomes. The ability of peripheral catheters to remain functional and in place without complications is crucial. While various clinical factors influence peripheral catheter performance, the composition and structure of peripheral catheters also affect their dwell time, which is defined as the duration at which the catheter remains functional after insertion. A study by McNeill et al. found that during the preintervention phase, about 62% of open-system peripheral catheters lost IV access within 36 hours, with less than 10% remaining functional beyond 72 hours. The dwell time of closed-system peripheral catheters with a securement device increased to up to 96 hours during the intervention period.8

DETAILED DESCRIPTION:
Peripheral catheters are the most frequently used medical devices in acute care settings, primarily for intravenous medication, fluid, and blood administration.1 However, their use is linked to various complications and risks, such as phlebitis, pain, infiltration, hematoma, occlusion, and more severe issues like bacteremia and sepsis.2 Studies indicate that the failure rate of peripheral catheters ranges between 35% and 50%, often due to dislodgment, infiltration, and other factors.2 These failures can lead to repeated venipunctures, increasing the risk of infection, pain, and potential damage to veins, all of which can impact patient comfort.

Advancements in the design and materials of peripheral catheters have improved their safety and comfort over time. These improvements include developing materials better suited for extended venous dwell time, mechanisms to prevent needle-related injuries, and securement devices, extension sets, stopcocks, and hubs. 3 The equipment needed for catheter insertion and maintenance varies, often consisting of multiple components that must be connected either before or after insertion. However, the manipulation of these components can introduce several issues. For instance, breaches in aseptic technique during this process can lead to the introduction of microbes into the patient's bloodstream, potentially causing insertion-related bacteremia. Previous studies have shown that Staphylococcus aureus is present in 7.6% to 23.5% of such cases.4,5 Catheter movement during manipulation can also result in dislodgment and loss of venous access. 3 One type of peripheral catheter, known as an open system, features a hub with an open end. These systems require additional components to complete the IV circuit, some of which are packaged separately. In open-system catheters, blood can flow out of the cannula and the open hub during venous access, leading to blood spillage and potential contamination. To address this, newer open-system catheters include features to prevent blood flow out of the hub after insertion, reducing the risk of blood spillage.

Another type of peripheral catheter is the closed system, which integrates an extension tube that contains blood flow within the circuit during cannulation. This design helps prevent blood spillage and needle-stick injuries. Closed-system peripheral catheters are self-contained units that do not require additional components for the IV circuit, reducing common points of contamination. Some closed-system peripheral catheters also include an integrated stabilisation platform to secure the catheter's position, which may help prevent dislodgment or injury to the vein.

Studies have shown that stabilisation devices are associated with fewer complications and lower failure rates in peripheral catheters.3,6,7 Although closed-system peripheral catheters offer potential advantages, such as reduced manipulation of components and minimised blood spillage, more research is needed to understand their impact on outcomes. The ability of peripheral catheters to remain functional and in place without complications is crucial. While various clinical factors influence peripheral catheter performance, the composition and structure of peripheral catheters also affect their dwell time, which is defined as the duration at which the catheter remains functional after insertion. A study by McNeill et al. found that during the preintervention phase, about 62% of open-system peripheral catheters lost IV access within 36 hours, with less than 10% remaining functional beyond 72 hours. The dwell time of closed-system peripheral catheters with a securement device increased to up to 96 hours during the intervention period.8

ELIGIBILITY:
Inclusion Criteria:

1. All patients admitted to the intensive care unit and requiring intravenous cannulation for dispensing drugs

Exclusion Criteria:

1. Patients with peripheral catheters inserted elsewhere before RICU admission 2 . Central venous catheters or other central vascular access devices 3. those with RICU stay < 24 hours will be excluded from the study 4. Pregnancy

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dwell time | 28 days
  Time till cannula is used for dispensing drugs
Dwell time | 28 days
  The time for which intravenous cannula is kept for dispensing drugs

SECONDARY OUTCOMES:
Catheter-related complications | 28 days
  Complications attributed to the intravenous cannula

CONTACTS AND LOCATIONS:
Overall Officials: Inderpaul S Sehgal, DM, Principal Investigator — PGIMER, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on reasonable request to the PI. The IPD will be shared for academic purposes and if the protocol is approved by the PI's IEC